CLINICAL TRIAL: NCT00612885
Title: Post Marketing Surveillance to Assess the Safety and Efficacy of Mobic® (Meloxicam) Intramuscular Injection (7.5mg ~ 15mg, q.d.) up to 3 Days (in Case of Need for Prolonged Treatment, Switch to Mobic® Capsule Therapy Was Possible) in Korean Patients With Osteoarthritis and Rheumatoid Arthritis (KFDA Regulatory Requirement PMS)
Brief Title: Safety and Efficacy of Mobic Inj. (Meloxicam) for the Patients With OA or RA: Observational Study
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Other Study IDs: 107.270
Record Dates: First submitted 2008-01-30; First posted 2008-02-12 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Osteoarthritis; Arthritis, Rheumatoid
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

SUMMARY:
The main objective of this PMS study was to monitor and assess the safety of Mobic® intramuscular injection (7.5mg ~ 15mg, q.d.) up to 3 days (in case of need for prolonged treatment, switch to Mobic® capsule therapy was possible) in Korean patients with osteoarthritis and rheumatoid arthritis.

ELIGIBILITY:
INCLUSION CRITERIA:

diagnosed as osteoarthritis and rheumatoid arthritis

EXCLUSION CRITERIA:

1. Known hypersensitivity to meloxicam
2. Cross hypersensitivity to aspirin and other non-steroidal anti-inflammatory drugs
3. Symptoms of asthma, rhinitis, angioneurotic edema, or urticaria following the administration of aspirin or other NSAIDs
4. Active peptic ulceration
5. Severe hepatic failure.
6. Non-dialysed severe renal insufficiency
7. Children and adolescents aged 15 years or less
8. Pregnancy or breastfeeding

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2004-03; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Efficacy assessment by the treating physician | up to 3 day
Combined efficacy, safety and tolerability assessment by the treating physician | up tp 3 day
Incidence of adverse events | up tp 3 day

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Korea Ltd.
Locations (11):
- South Korea (11):
  - Boehringer Ingelheim Investigational Site, Busan
  - Boehringer Ingelheim Investigational Site, Daegu
  - Boehringer Ingelheim Investigational Site, Daejeon
  - Boehringer Ingelheim Investigational Site, Gangwondo
  - Boehringer Ingelheim Investigational Site, Gwangju
  - Boehringer Ingelheim Investigational Site, Gyeongbuk
  - Boehringer Ingelheim Investigational Site, Gyeonggido
  - Boehringer Ingelheim Investigational Site, Gyeongnam
  - Boehringer Ingelheim Investigational Site, Jeonnam
  - Boehringer Ingelheim Investigational Site, Jungbuk
  - Boehringer Ingelheim Investigational Site, Seoul